CLINICAL TRIAL: NCT05873296
Title: Impact of Health Education on Lifestyle for Women With Breast Cancer: Health Education
Brief Title: Health Education for Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Maranhao (Other)
Responsible Party: Principal Investigator, Andréa Dias Reis, Principal Investigator, Federal University of Maranhao
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UFMA
Record Dates: First submitted 2023-03-22; First posted 2023-05-24 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Female
Keywords: Breast Neoplasms; Sedentary Behavior; Lifestyle; Health Education
MeSH Terms: conditions — Breast Neoplasms; Sedentary Behavior; Health Education

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Education (Experimental): Group of women being treated for breast cancer
  Interventions: Behavioral: Health Education
- usual care (No Intervention): Group of women who will remain in usual care

INTERVENTIONS:
Behavioral: Health Education — The intervention will last for 12 weeks, a health education program (face-to-face meetings and information in social networks).
  Arms: Health Education

SUMMARY:
The sedentary lifestyle in women with breast cancer generates a problem for public health. An alternative that has been used to reduce sedentary behavior are interventions with the use of information technology, as well as projects with health education can cause lifestyle changes. However, little is known about the effect of these interventions on self-awareness and self-care in women with breast cancer. This aim of study is evaluate the effect of health education on sedentary behavior, lifestyle, physical activity level, nutrition, self-esteem, anxiety and depression, quality of life, pain, functional capacity, and strength in women with breast cancer. This is a study the 12 weeks, with patients being treated for breast cancer, distributed for two groups: Group Health Education Recommendations and Control Group.

DETAILED DESCRIPTION:
This is a clinical trial with patients being treated for breast cancer, the sample will be randomly distributed into two groups: Group Health Education Recommendations (GRES) and Control Group (CG), which will remain in usual care. The intervention will last for 12 weeks, where GRES will receive health education recommendations in person and via social media. The endpoints of this study are sedentary behavior, lifestyle, physical activity level, nutrition, self-esteem, anxiety and depression, quality of life, pain, functional capacity, and strength. Evaluations will be performed at baseline, after 6 weeks, and after 12 weeks. Data will be analyzed by multivariate, comparing the effects of group, time, and interaction in SPSS software version 24.0, with α=5%.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older;
* Diagnosed with breast cancer;
* Ongoing breast cancer treatment (chemotherapy, radiotherapy and/or hormone therapy);
* Have daily access to a smartphone.

Exclusion Criteria:

* Women having another type of cancer;
* Perform physical training for three months before the intervention;
* Has medical contraindication to perform any type of physical activity;
* Have filled in yes on the PAR-Q and medical contraindication;
* Without cognitive conditions to use a smartphone or answer questionnaires;
* Illiterate women.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Life habits | Change from baseline, 6 weeks Life habits at 12 weeks
  Lifestyle will be evaluated by Individual Lifestyle Profile Questionnaire (score 0 to 3 - higher score is better)

SECONDARY OUTCOMES:
Body composition (lean mass, fat mass) | Change from baseline, 6 weeks Body composition at 12 weeks
  Body Composition will be evaluated by Sanny Tetrapolar Bioimpedance (Model 1011)
Sitting time | Change from baseline, 6 weeks Sitting time at 12 weeks
  Sedentary behavior will be evaluated by triaxial accelerometers motion sensor Actigraph GT3X model
Time and level the physical activity | Change from baseline, 6 weeks Time and level the physical activity at 12 weeks
  Physical activity level will be evaluated by triaxial accelerometers motion sensor Actigraph, GT3X model.
Level the self-esteem | Change from baseline, 6 weeks Level the self-esteem at 12 weeks
  Self-esteem will be evaluated by Rosenberg Self-Esteem Scale (score 1 to 4 - higher score is better and worse outcome, depends on the question)
Dimensions the quality of Life from cancer | Change from baseline, 6 weeks Dimensions the quality of Life at 12 weeks
  Quality of Life will be evaluated by European Organization for Research and Treatment of Cancer Quality of Life Questionnarie - 30 questions (score 1 to 4 - higher score is worse outcome)
Dimensions the quality of Life from breast cancer | Change from baseline, 6 weeks Dimensions the quality of Life at 12 weeks
  Quality of Life will be evaluated by European Organization for Research and Treatment of Cancer Quality of Life Questionnarie - 23 questions (score 1 to 4 - higher score is worse outcome)
Level the pain | Change from baseline, 6 weeks Level the pain at 12 weeks
  Pain will be evaluated by Brief Pain Inventory (score 1 to 10 - higher score is worse outcome)
Eating habits | Change from baseline, 6 weeks Eating habits at 12 weeks
  Eating behavior will be evaluated by (score 1 to 4 - higher score is better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Andréa D Reis, Principal Investigator — Federal University of Maranhão
Locations (1):
- Andréa Dias Reis, São Luís, Maranhão, Brazil

REFERENCES:
- See also: AMERICAN CANCER SOCIETY — https://www.cancer.org/cancer/breast-cancer/treatment.html
- See also: World Health Organization — https://www.who.int/pt/news/item/03-02-2021-breast-cancer-now-most-common-form-of-cancer-who-taking-action